CLINICAL TRIAL: NCT04154553
Title: Pharmacogenetic Testing of Patients With Unwanted Adverse Drug Reactions or Therapy Failure
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Toppharm Apotheke Hersberger, Spalenberg 41, CH-4051 Basel (Unknown); Universitätskinderspital Zürich, Lenggstrasse 30, 8008 Zürich (Unknown); Institut für Spitalpharmazie, Solothurner Spitäler AG, Baslerstrasse 150, 4600 Olten (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019-01452; ex19Hersberger
Record Dates: First submitted 2019-10-31; First posted 2019-11-06 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Adverse Drug Reaction; Therapy Failure
Keywords: pharmacogenetics; single nucleotide polymorphism; absorption, distribution, metabolism and excretion (ADME); genotyping; pharmacogenetic testing
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The buccal swab and the extracted DNA are destroyed after two to three weeks after the accomplished labor analysis. The coded ethylenediaminetetraacetic acid (EDTA) blood samples will be stored at -80°C in the Biobank of Biopharmacy Laboratory until further use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Buccal swab — Pharmacogenetic panel testing is conducted by Stratipharm with the DNA of the buccal swab. TaqMan® polymerase chain reaction is proceeded to express the genetic information. Stratipharm is a product offered by Humatrix Aktiengesellschaft (AG). It consists of a laboratory analysis of approximately 100 pharmacological relevant genetic variations (polymorphisms) in over 30 different genes, which code for transport proteins, metabolizing enzymes, or drug targets.
Diagnostic Test: EDTA Blood sample (4.9mL) — Genetic testing of potentially relevant genetic variants using the DNA extracted from the EDTA blood sample.
Diagnostic Test: Serum sample (7.5mL) — blood sample to determine the actual levels of the compound in patients on medication assumed to be associated to an observed ADR (phenotype).
Other: communication of test results — Certified study pharmacist evaluates and communicates clinically relevant test results to the subject and to the responsible physician
Other: unstructured interview — One and six months after the communication of test results, the study center will make a phone call to the patient for an unstructured interview in order to gather information about potential outcomes

SUMMARY:
Genetic makeup of a patient influences the efficacy and safety profile of a drug. This study is to summarize individual cases, where Pharmacogenetics (PGx) has been applied during pharmaceutical care. The primary objective is the compilation of case reports, where pharmacogenetic testing is applied to determine the hereditable component of the patient's susceptibility to experience therapy failure and/or adverse drug reactions. The experience with the compiled cases will be basis for the development of a reliable standard of procedure for pharmacogenetic testing in the community pharmacy. The cases will be supplemented with information on additional Parameters reported in the literature to affect efficacy or safety of the respective drug.

DETAILED DESCRIPTION:
Genetic makeup of a patient influences the efficacy and safety profile of a drug. This study is to summarize individual cases, where Pharmacogenetics (PGx) has been applied during pharmaceutical care. Health-related data of patients experiencing therapy failure (TF) or adverse drug reaction (ADR) is collected and will then be supplemented with pharmacogenetic testing during pharmaceutical care in a study pharmacy. The patient data (diagnoses, medications and results of pharmacogenetic testing) is harmonized in order to generate a compilation of case reports. The primary objective is the compilation of case reports, where pharmacogenetic testing is applied to determine the hereditable component of the patient's susceptibility to experience therapy failure and/or adverse drug reactions. The experience with the compiled cases will be basis for the development of a reliable standard of procedure for pharmacogenetic testing in the community pharmacy. The cases will be supplemented with information on additional Parameters reported in the literature to affect efficacy or safety of the respective drug.

ELIGIBILITY:
Inclusion Criteria:

* New medication with known PGx association (preemptive)
* Current medication with observation of adverse drug reactions probably linked to drugs with known PGx association (reactive)
* Current medication with observation of therapy failure probably linked to drugs with known PGx association (reactive)
* Current and/or new medication and a family history of adverse drug reactions/therapy failure probably linked to drugs with known PGx association
* Signed informed consent; for patients < 14 years, the legal representative needs to sign the informed consent

Exclusion Criteria:

* Insufficient German knowledge
* Not able to personally visit to the study pharmacy

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The patient population are patients experiencing TF and/or ADRs with substances known to be affected by genetic variants that influence their drug metabolism (pharmacokinetics) and/or the activity of the drug target (pharmacodynamics).
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
pharmacogenetic profile | single time point assessment at Baseline (=Day 0)
  genotyping by laboratory analysis of approximately 100 pharmacological relevant genetic variations (polymorphisms) in over 30 different genes

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Hersberger, Prof. Dr., Study Chair — Pharmaceutical Care Research Group; Department of Pharmaceutical Sciences, University Basel; Samuel Allemann, Prof. Dr., Principal Investigator — Pharmaceutical Care Research Group; Department of Pharmaceutical Sciences, University Basel
Locations (1):
- Department of Pharmaceutical Sciences, University Basel, Basel, Switzerland